CLINICAL TRIAL: NCT06926920
Title: A Phase 1/2, Open-label Study of Sacituzumab Govitecan Administered at an Alternative Dose and Schedule in Participants With Advanced Triple-Negative Breast Cancer
Brief Title: A Study of Sacituzumab Govitecan Given at an Alternative Dose and Schedule in Participants With Advanced Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-576-7321; 2024-519124-25 (Other: European Medicines Agency); 2024-519124-25 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): Participants will receive SG until progressive disease (PD), death, unacceptable toxicity, or another treatment discontinuation criterion is met.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG)
- Phase 2: Expansion (Experimental): Participants will receive SG until PD, death, unacceptable toxicity, or another treatment discontinuation criterion is met.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG)

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy (SG) — Administered intravenously
  Other Names: GS-0132; Trodelvy

SUMMARY:
The goal of this clinical study is to learn more about the study drug sacituzumab govitecan-hziy (SG) given at an alternative dose and schedule, in participants with triple-negative breast cancer (TNBC).

The primary objectives of this study are to assess the safety and tolerability of SG given at alternate dose and schedule, to assess the effect on objective response rate (ORR) and progression-free survival (PFS).

DETAILED DESCRIPTION:
Phase 1 of this study will evaluate the preliminary safety, tolerability, pharmacokinetics (PK), and efficacy of SG. Phase 2 expansion of this study will further evaluate the safety, efficacy, and PK of SG.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals assigned male or female at birth, 18 years of age or older, able to understand and give written informed consent.
* Histologically or cytologically locally confirmed TNBC.
* Phase 1: Individuals with unresectable, locally advanced or metastatic TNBC who are refractory to or relapsed after at least one prior standard-of-care chemotherapy regimen or systemic therapy given for locally advanced or metastatic disease.
* Phase 2: Individuals with unresectable, locally advanced or metastatic TNBC who have not received previous systemic therapy for advanced disease.
* Phase 2: Tumors must be PD-L1 negative, defined as tumor PD-L1 combined positive score (CPS) < 10 using the PD-L1 immunohistochemistry (IHC) 22C3 assay. Alternatively, individuals with tumor CPS ≥ 10 will be eligible if they received an anti-PD-(L)1 agent (ie, checkpoint inhibitor) in the adjuvant or neoadjuvant setting or if they cannot be treated with an anti-PD-(L)1 agent. due to a comorbidity.
* Uridine diphosphate glucuronosyltransferase 1A1 (UGT1A1) genotype status.

During Phase 1 safety run-in, individuals must be UGT1A1 wild-type.

After Phase 1 safety run-in, individuals with any UGT1A1 genotype may be eligible.

* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) according to RECIST Version 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate hematologic counts within 2 weeks prior to enrollment.
* Adequate hepatic and renal function.

Key Exclusion Criteria:

* Prior treatment with a topoisomerase 1 inhibitor or antibody-drug conjugate (ADC) containing a topoisomerase inhibitor.
* Prior treatment with a trophoblast cell-surface antigen 2 (Trop-2)-directed ADC.

Note: Other protocol defined Inclusion/Exclusion criteria will apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Percentage of Participants Experiencing Dose-Limiting Toxicities (DLTs) | First dose up to 28 days
Phase 1 and 2: Percentages of Participants Experiencing Adverse Events (AEs) | First dose up to 30 days post last dose (Up to 3 years)
Phases 1 and 2: Percentages of Participants Experiencing Laboratory Abnormalities | First dose up to 30 days post last dose (Up to 3 years).
Phases 1 and 2: Percentages of Participants Experiencing AEs Leading to Dose Reductions, Dose Interruptions, and Treatment Discontinuations | First dose up to 30 days post last dose (Up to 3 years).
Phases 1 and 2: Objective Response Rate (ORR) | Up to 9 months
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) that is confirmed at least 4 weeks after initial documentation of response as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Phase 2: Progression-Free Survival (PFS) | Up to 9 months
  PFS is defined as the time from the date of the first SG dose until the date of progressive disease (PD) as assessed by the investigator according to RECIST Version 1.1, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Phases 1 and 2: Serum Concentrations of SG | Up to End of Treatment (3 years)
Phase 1 and 2: Percentage of Participants who Develop Antidrug Antibodies (ADAs) Against SG | First dose up to 30 days post last dose (Up to 3 years).
Phase 2: Duration of Response (DOR) | First dose up to 30 days post last dose (Up to 3 years).
  DOR is defined as the time from the first documentation of CR or PR to the first documentation of PD as assessed by the investigator according to RECIST Version 1.1, or death from any cause, whichever occurs first.
Phase 2: Disease Control Rate (DCR) | Up to 9 months
  DCR is defined as the proportion of participants who achieve CR, PR, or stable disease as assessed by the investigator according to RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (16):
- United States (9):
  - Los Angeles Cancer Network (LACN) - Good Sam, Los Angeles, California
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - The University of Kansas Hospital, Westwood, Kansas
  - Siteman Cancer Center, St Louis, Missouri
  - West Cancer Centre, Germantown, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology - DFW, Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Australia (3):
  - St. Vincent's Hospital - Kinghorn Cancer Center, Darlinghurst, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - John Flynn Private Hospital, Tugun, Queensland
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06926920